CLINICAL TRIAL: NCT00315965
Title: Development of a New Method for Steady-State Measurement of NO Lung Diffusing Capacity in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ESNOD-01
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2007-05

CONDITIONS: Pulmonary Diffusing Capacity
Keywords: Diffusion; Membrane diffusing capacity; Alveolar capillary gas diffusion; Transfer factor; Nitric oxide diffusion
MeSH Terms: interventions — Nitric Oxide; Carbon Monoxide; Helium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nitric oxide, Carbon monoxide, Helium

SUMMARY:
Using a rapidly responding nitric oxide analyzer in a new developed modular lung-function-setup we are going to measure steady-state NO diffusing capacity in 107 healthy subjects (age 6-45 years). The results will be compared to those measured by using carbon monoxide single-breath estimates. We like to show that the new method is sufficient to measure exactly lung diffusion capacity in this collective.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Lung function testing possible
* Written consent

Exclusion Criteria:

* Pulmonary, neuromuscular, cardiovascular, endocrinological illness
* Pregnancy
* Abuse of nicotine, alcohol, drugs during the last two years

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 107 (Estimated)
Dates: Start 2006-07; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
TLNOss
TLCOsb

SECONDARY OUTCOMES:
Breathing frequency
tidal volume
functional residual capacity
airway resistance
lung clearance index
forced expiratory volume in one second
vital capacity
total lung capacity

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Pantalitschka, MD, Principal Investigator — University Hospital Tuebingen, Germany
Locations (1):
- University children´s hospital, Tübingen, Germany